CLINICAL TRIAL: NCT03588611
Title: The Noninferiority and Safety of Bivalirudin Between REDUCEd and Standard BOLUSin Percutaneous Coronary Intervention Patients Stratified by Renal Function
Brief Title: Reduce Bolus Injection of Bivalirudin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Han Yaling, MD (Other)
Responsible Party: Sponsor-Investigator, Han Yaling, MD, The noninferiority and safety of bivalirudin between REDUCEd and standard BOLUSin percutaneous coronary intervention patients stratified by renal function, Shenyang Northern Hospital
Organization: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RE-20180628
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Acute Coronary Syndrome
Keywords: bivalirudin; bolus injection; activated clotting time; Renal insufficiency
MeSH Terms: conditions — Acute Coronary Syndrome; Renal Insufficiency | interventions — bivalirudin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low dose group with eGFR ≥60ml/min (Experimental): This arm, we will choose the patients who's eGFR ≥60ml/min and reduce the bivalirudin bolus injection dose to 80% of the standard dose in clinical practice, and we will adjuste the bivalirudin maintenance dose and rate according to the ACT time during surgery to reduce the ACT value caused by the bolus injection.
  Interventions: Drug: Bivalirudin
- Standard dose group with eGFR ≥ 60ml/min (Active Comparator): This arm, we will choose the patients who's eGFR ≥60ml/min and use the standard dose in clinical practice, and we will adjuste the bivalirudin maintenance dose and rate according to the ACT time during surgery .
  Interventions: Drug: Bivalirudin
- Standard dose group with eGFR <60ml/min (Active Comparator): This arm, we will choose the patients who's eGFR <60ml/min and use the standard dose in clinical practice, and we will adjuste the bivalirudin maintenance dose and rate according to the ACT time during surgery .
  Interventions: Drug: Bivalirudin
- Low dose group with eGFR <60ml/min (Experimental): This arm, we will choose the patients who's eGFR <60ml/min and reduce the bivalirudin bolus injection dose to 80% of the standard dose in clinical practice, and we will adjuste the bivalirudin maintenance dose and rate according to the ACT time during surgery to reduce the ACT value caused by the bolus injection.
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Bivalirudin — 0.75mg/kg+ 1.75 mg/kg▪h for the duration of PCI;
  Arms: Standard dose group with eGFR <60ml/min; Standard dose group with eGFR ≥ 60ml/min
Drug: Bivalirudin — 0.6mg/kg+ 1.75 mg/kg▪h for the duration of PCI;
  Arms: Low dose group with eGFR <60ml/min; Low dose group with eGFR ≥60ml/min

SUMMARY:
There are fewer studies on the bleeding risk of the currently administered bivalirudin bolus injection dose and the safety of bivalirudin in patients with CKD. A non-inferiority, randomized, stratified controlled trial study has been conducted to evaluate the non-inferiority and safety of the low dose (80%) bolus injections of bivalirudin in patients with or without CKD.This study will provide a safe, effective and economical anticoagulation strategy.

ELIGIBILITY:
Inclusion Criteria:

* 1 Age 18 to 80 years old; 2 Medically judge to require coronary angiography; 3 Patients agree to use bivalirudin 4 Patients signe informed consent.

Exclusion Criteria:

* 1.Cardiogenic shock; 2.Thrombolytic therapy administered before randomization or any anticoagulant administered within 48 hours of randomization; 3.Active or recent major bleeding or bleeding predisposition; 4.Major surgery within 1 month; 5.Clinical syndrome suspicious for aortic dissection, pericarditis, or endocarditis; blood pressure higher than 180/110 mm Hg; 6.Known hemoglobin less than 10 g/dL,platelet count less than 100 × 109/L, aminotransferase level greater than 3 × the upper limit of normal; 7.History of heparin-induced thrombocytopenia; 8.Ellergy to any of the study drugs or devices; 9.Eregnancy or lactation; 10.Any condition making PCI unsuitable or that might interfere with study adherence; 11.Patient unwilling or unable to provide written informed consent 12. Researchers think it is not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
The area under the curve of the ACT values for both groups | During operation
  We will record the ACT values of 0 min, 5 min, 10 min, and 30 min after bolus injection of bivalirudin in patients undergoing PCI,and the area of the closed pattern under the curve will be calculated, and the anticoagulant effect of bivalirudin will be evaluated by the area under the ACT line.

SECONDARY OUTCOMES:
Incidence of bleeding and ischaemic events during hospitalization after surgery . | In hospital
  Bleeding events are defined as BARC grade 1-5. Ischemic events are defined as stroke, nonfatal myocardial reinfarction, ischemic-driven target vessel revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Hu Q, Han YL, Zhou TN, Wang XZ, Zhang QY. Efficacy and Safety of the Reduced Bivalirudin in Patients Undergoing Coronary Angiography or Percutaneous Coronary Intervention Stratified by Renal Function (REDUCE BOLUS): A Single-Blind, Stratified Randomized, Non-inferiority Trial. Front Cardiovasc Med. 2022 Apr 25;9:864048. doi: 10.3389/fcvm.2022.864048. eCollection 2022. PMID 35548446